CLINICAL TRIAL: NCT02188836
Title: Electromagnetic Stimulation as Coadjuvant in the Healing of Diaphyseal Femoral Fractures: a Randomized Controlled Trial
Brief Title: Electromagnetic Stimulation as Coadjuvant in the Healing of Diaphyseal Femoral Fractures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Principal Investigator, Juan Pablo Martinez, Medical doctor, Fundacion Clinica Valle del Lili
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FemurEMG
Record Dates: First submitted 2014-06-27; First posted 2014-07-14 (Estimated); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Fracture, Closed, Comminuted, Healing
MeSH Terms: conditions — Fractures, Bone; Fractures, Comminuted

STUDY DESIGN:
Intervention Model Description: Electromagnetic device
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sham electromagnetic device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electromagnetic device (Experimental): The electromagnetic stimulation was performed by using a device capable of generating an electromagnetic field around the fracture site. This was applied once a day, one hour for 8 weeks.
  Interventions: Device: Electromagnetic stimulation
- Placebo device (Placebo Comparator): A device with the same characteristics to the real device, except for the generation of the electromagnetic stimulation. It generates sham stimulation.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Electromagnetic stimulation — Electromagnetic stimulation with a new device produced by the investigators for this study.
  Other Names: "Consolidator"
  Arms: Electromagnetic device
Device: Sham stimulation — This is a device that look exactly the same to the electrostimulation device, but that does not generate the electromagnetic field. It is a placebo device.
  Arms: Placebo device

SUMMARY:
This study specifically evaluates the effects of electromagnetic stimulation for diaphyseal femur fractures using a device developed by the investigators.

The hypothesis is that patients with femoral diaphysis treated with the electromagnetic stimulation have less non-union after six months than patients treated with a placebo device.

DETAILED DESCRIPTION:
The inclusion criteria were: patients of any sex, age between 18 and 60 years, with a closed fracture in their femoral diaphysis or an open fracture secondary to a low-speed bullet; treated with open or closed reduction and intramedullary reamed blocked nail.

Patients were excluded if they had a pathological fracture, an open fracture from another etiology, or if they were treated after 10 days from the day of fracture.

64 patients were included.

Randomization took place six weeks after fracture day, allocating participants to either one of two groups: group A (electromagnetic stimulation) or group B (placebo).

Each group had a device exactly the same. Patients used the device during one hour every day for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any sex,
* age between 18 and 60 years, with a closed fracture in their femoral diaphysis or an open fracture secondary to a low-speed bullet;
* treated with open or closed reduction and intramedullary reamed blocked nail.

Exclusion Criteria:

* Patients were excluded if they had a pathological fracture,
* an open fracture from another etiology, or if they were treated after 10 days from the day of fracture.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2008-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Fracture healing | up to 18 weerks
  Percentage (%) of patients with their fracture healed six months after the fracture day and 18 weeks after treatment began.

SECONDARY OUTCOMES:
Infection | 6 months
  Percentage (%) in each arm which may present an infection.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Martinez, MD, Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundacion Valle del Lili, Cali, Valle del Cauca Department, Colombia